CLINICAL TRIAL: NCT06431867
Title: A Qualitative Exploration of Older Women and Primary Healthcare Professional Experiences to Guide Improvements in Osteoporosis Care
Brief Title: Primary Care Management of Osteoporosis in Older Women
Status: Recruiting | Type: Observational
Sponsor: Bradford Institute for Health Research (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Principal Investigator, Anne Heaven, Research Programme Manager, Bradford Institute for Health Research
Other Study IDs: BTHFT2918; NIHR205378 (Other Grant/Funding Number: National Institute for Health and Care Research (NIHR))
Record Dates: First submitted 2024-05-22; First posted 2024-05-29 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Osteoporosis
Keywords: women; older; primary-care
MeSH Terms: conditions — Osteoporosis | interventions — Guidelines as Topic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Older women: Women aged 70 years and older with a diagnosis of osteoporosis
  Interventions: Other: Guidelines for primary care management of osteoporosis
- Primary healthcare professionals: Any healthcare professional working in a primary care setting e.g. general practitioner, pharmacist, physiotherapist
  Interventions: Other: Guidelines for primary care management of osteoporosis

INTERVENTIONS:
Other: Guidelines for primary care management of osteoporosis — All usual care of osteoporosis in primary care

SUMMARY:
The Investigators aim to improve primary-care for older women with osteoporosis.

Older women they spoke with previously felt unseen, unimportant, unheard and uninformed. These women felt that bone/joint health was an important issue for women aged 70+. Osteoporosis is a disease that makes bones more breakable and can lead to significant pain, disability and death, costing approximately £4.4 billion a year in the United Kingdom.

Women are four times more likely to have osteoporosis than men and suffer fractures earlier. Osteoporosis care is poor in primary care even though good guidelines are available.

The Investigators will work with older women and healthcare professionals to help guide the research. They have already looked at published research and will build on this. They will identify what is important for both older women and professionals to inform the first interview questions. The Investigators will ask older women and healthcare professionals about the diagnosis and treatment of osteoporosis. They will also ask them how they manage osteoporosis as a patient or care provider.

At regular intervals, the Investigators will look at the interview findings first and then share their thoughts with older women and professionals. Together they will explore what the interviews mean. These discussions may change the questions asked and who is interviewed next.

The Investigators will combine all the information from interviews to identify what works well and less well in osteoporosis care. They will check these findings against the guidelines. They will continue to work with older women and healthcare professionals to develop recommendations for improving care. The Investigators will also identify areas of further work.

They will share recommendations with healthcare commissioners and produce a summary for a variety of professional networks. They will also publish papers in journals aimed at healthcare professionals and produce a summary document and advice for older women to use.

DETAILED DESCRIPTION:
RESEARCH QUESTION How can older women and primary healthcare professionals be empowered to improve osteoporosis care?

BACKGROUND The Women's Health Strategy for England highlights the lack of focus on older women's needs and experiences. The Investigators talked to 32 older women across five public engagement workshops. These women felt unseen, unimportant, unheard and uninformed. They also felt bone/joint health and osteoporosis were important issues for older women (aged 70+). Osteoporosis leads to around 180,000 fractures per year causing significant pain, disability and death. The related cost, in the United Kingdom, is estimated at £4.4 billion a year. Women are four times more likely to suffer with osteoporosis than men and tend to suffer fractures earlier. Despite comprehensive guidelines being available, evidence suggests that osteoporosis care is lacking in primary care.

AIMS AND OBJECTIVES To develop strategies to improve osteoporosis care using insights from the experience of primary healthcare professionals and older women.

METHODS Ethnographic meta-analysis literature review, in-depth interviews and co-production workshops. An information specialist will update the preliminary literature review. The Investigators will synthesise evidence from older women and healthcare professionals to identify new theoretical constructs. Findings will be reviewed in co-production workshops and used to focus initial lines of enquiry. The Investigators will purposively sample 30 older women, from across England, aged 70+ to interview. They will also elicit the views of healthcare professionals in primary care. Interviews will explore the process of diagnosis, treatment and management of osteoporosis. Information from interviews will initially be reviewed by the Investigators.

Following a Constructivist Grounded Theory approach, the Investigators will take initial findings to co-production workshops on a regular basis throughout fieldwork. Workshops will facilitate iterative analysis and identify theoretical sampling gaps. This process may change the types of questions asked or who is interviewed. The Investigators will combine information from all interviews to identify barriers and facilitators for older women's osteoporosis care, and cross-reference this with existing guidelines. Professional 'expert witnesses' will join the workshops when required. Finally, recommendations for improving osteoporosis care will be co-produced . Areas of further work that would improve osteoporosis care in the future will also be identified.

PATIENT AND PUBLIC INVOLVEMENT Lay members will be involved in co-production workshops throughout the research. The Investigators will also work with an expert patient co-applicant in overall management of the project.

TIMELINES FOR DELIVERY Following 3 months of pre-award set-up, the Investigators will conduct the literature review and develop the interview schedule in months 1-3. Interviews and workshops will happen in months 4-11. A final analysis and report will be available in month 18.

IMPACT AND DISSEMINATION Findings will be sent to Integrated Care Boards responsible for local commissioning to facilitate 'better fit' services. The Investigators will also produce dissemination products for wide distribution through a variety of professional networks. Academic papers will be published in journals targeted at healthcare professionals. Summary information and advice, for older women, will be disseminated via national and community networks and presentations nationwide. These outputs will be aimed at supporting successful implementation of the All Party Parliamentary Group recommendations for better diagnosis, treatment and management.

ELIGIBILITY:
Inclusion Criteria

Older women:

* Osteoporosis diagnosis - either self-reported following a clinical diagnosis or taken from the patient's medical record in the case of the Community Ageing Research 75+ (CARE75+) cohort and Fracture Liaison Service (FLS) patients.
* Aged 70 years or older to align with the recommendation from our preliminary engagement work.
* Community dwelling.

Healthcare professionals:

• Working in the National Health Service (NHS) in England to align with the participant sample.

Exclusion criteria

Older women:

* Aged under 70 years.
* Lacks capacity to consent to participate in research.
* Resident in a care home - care home residents are likely to need different types of interventions than community dwelling older women as there are organisational considerations.
* Member of the co-production workshop.

Healthcare professionals:

* Not performing any NHS work.
* < 12 months in NHS practice.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Thirty women with a diagnosis of osteoporosis aged 70 years and older. The Investigators will purposively sample for maximum variation to ensure inclusion of people from a range of living circumstances, from a mixture of urban and rural locations and spanning the least deprived and most deprived locations (identified from Index of Multiple Deprivation (IMD) deciles based on postcode areas). Interview findings will be reviewed on a regular basis during the co-production workshops and adjusted as necessary to follow emergent leads.
  Thirty healthcare professionals using a purposive sample based on gender, number of years qualified and IMD score of practice catchment.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-09-16 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Questionnaire | September 2025
  Constructivist grounded theory about how osteoporosis in older women is treated and managed in primary care

CONTACTS AND LOCATIONS:
Overall Officials: Anne Heaven, MPhil, Principal Investigator — Bradford Institute for Health Research
Locations (1):
- Bradford Institute for Health Research, Bradford, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
All external data requests will be reviewed by the Project Management Group. Permission to access anonymised data will be subject to a data sharing agreement. Participants will be asked to explicitly consent to secondary data analysis - this will be optional.

REFERENCES:
- See also: Organisational website — http://ageingstrokeresearch.org/